CLINICAL TRIAL: NCT06459089
Title: The Effects of Familiar Toy and Parental Presence on Perioperative Pediatric Anxiety
Brief Title: The Effects of Familiar Toy and Parental Presence Combination on Perioperative Pediatric Anxiety
Status: Completed | Type: Observational
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 01-2024/13
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Perioperative Anxiety; Emergence Delirium
Keywords: Anxiety State; Familiar Toy; Child Behavior
MeSH Terms: conditions — Emergence Delirium; Anxiety Disorders; Child Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group1: The children will select the parent who acoompany theim during anesthesia induction
  Interventions: Behavioral: Selection of the parent according to children preference
- Group 2: The children will select the parent who accompany them dring anesthesia induction and bring their favorite toy also to the operating room.
  Interventions: Behavioral: Selection of the parent according to children preference; Behavioral: Bringing the favorite toy of the children that will accompany the child during their perioperative period

INTERVENTIONS:
Behavioral: Selection of the parent according to children preference — The children will select the parent who will accompany them during the anesthesia induction
Behavioral: Bringing the favorite toy of the children that will accompany the child during their perioperative period — The children will bring tiheir favorite toy that will accompany them during their perioperative period
  Groups: Group 2

SUMMARY:
This study will evaluate the effect of presence of favorite toy and parent during perioperative period on pediatric anxiety and emergence delirium. Half of the patients patients will be accompanied with their ownselected parent and the other half will be accompanied with their favorite toy in addition to their own selected parent.

DETAILED DESCRIPTION:
To reduce the incidence of preoperative anxiety in children, anesthesiologists have used a number of prevention strategies, including sedative premedication, parental presence during anesthetic induction, behavioral preparation programs, music therapy, hypnosis, and acupuncture.One of these distraction tool is familiar toy, children may also be comforted by familiar toys. Therefore, parent presence during perioperative period or playing with a favorite toy seems likely to alleviate preoperative anxiety in children. Until now, combination of these two method to reduce anxiety is not observed in literature. Then, the aim of this observational study is to evaluate the effect of both presence of favorite toy and parental presence compare to only parental presence during perioperative period on anxiety and emergence delirium in patients undergoing ambulatory surgery in our hospital's otorhinolaryngology department.

ELIGIBILITY:
Inclusion Criteria:

Patients with ASA 1 and 2, Those who have the ability to speak and obey commands will be included.

Exclusion Criteria:

Mentally challenged Deaf Child Cerebral Palsy Premedicated Child Language Problem Unco-operative Previous surgery or anesthesia history

Ages: 5 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: 100 child patients between the ages of 5-12 who will undergo ENT surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Modified Yale Preoperative Anxiety Scale (mYPAS) of the children undergoing elective surgery under general anesthesia. | Perioperative period
  The mYPAS will be used to evaluate the anxiety level of children. The mYPAS is an observational measure of preoperative anxiety consisting of 27 items in 5 domains (activity, emotional expressivity, state of arousal, vocalization, and use of parents). The adjusted mYPAS total score ranges from 22.9 to 100, with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Evaluation with Pediatric Anesthesia Emergence Delirium Scale (PAED) in the postoperative waiting room | Postoperative 1st day
  Incidence of post-anesthesia and postoperative delirium Discordant behaviors assessed with Pediatric Anesthesia Emergence Delirium Scale (PAED) with five features, each scored using a 5-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Duran, MD, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)